CLINICAL TRIAL: NCT02002429
Title: Medial Branch Blocks vs. Intra-articular Injections: Randomized, Controlled Study Comparing Lumbar Facet Radiofrequency Denervation Using Diagnostic Injections.
Brief Title: Medial Branch Blocks vs. Intra-articular Injections: Randomized, Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00086597
Record Dates: First submitted 2013-12-01; First posted 2013-12-05 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Lumbar Facet Joint Pain; Low Back Pain
Keywords: Facet joint; Medial branch block; Radiofrequency denervation; Zygapophysial joint; Low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Injections, Intra-Articular; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intra-articular injection (Experimental): Intra-articular injection into the affected facet joint(s) with 0.5 ml of a 50:50 solution containing 10 mg of depo-methylprednisolone and 0.5% bupivacaine
  Interventions: Procedure: Intra-articular injection
- Medial branch block (Active Comparator): Medial branch blocks at the nerves that supply the affected facet joint(s) with 0.5 ml of a 50:50 solution containing 10 mg of depo-methylprednisolone and 0.5% bupivacaine
  Interventions: Procedure: Medial branch block
- Saline injection (Sham Comparator): Injection into the affected facet joint(s) with 0.5 ml of normal saline
  Interventions: Procedure: Saline injection

INTERVENTIONS:
Procedure: Intra-articular injection — Intra-articular injection into the affected facet joint(s) with 0.5 ml of a 50:50 solution containing 10 mg of depo-methylprednisolone and 0.5% bupivacaine. If the subject has a positive block a radiofrequency denervation will be performed at the affected joint.
  Arms: Intra-articular injection
Procedure: Medial branch block — Medial branch blocks at the nerves that supply the affected facet joint(s) with 0.5 ml of a 50:50 solution containing 10 mg of depo-methylprednisolone and 0.5% bupivacaine. If the subject has a positive block a radiofrequency denervation will be performed at the affected joint.
  Arms: Medial branch block
Procedure: Saline injection — Injection into the affected facet joint(s) with 0.5 ml of normal saline. All subjects in the group will receive radiofrequency denervation.
  Arms: Saline injection

SUMMARY:
Background: Facet interventions are the second most commonly performed procedure in pain clinics throughout the U.S, including in the military. Currently, there is no clear consensus regarding whether intra-articular (IA) blocks or medial branch blocks (facet joint nerve; MBB) are the best way to diagnose and treat facetogenic pain, or even whether or not to perform diagnostic/ prognostic blocks.

Hypothesis: IA blocks will provide better relief than MBB, but MBB may better select patients for radiofrequency denervation.

Purpose: Objective 1: Determine which "prognostic" block is the best predictor for RF denervation outcome; Objective 2: To determine whether adding steroids to IA or MBB may provide intermediate or long-term benefit to a subset of individuals.

Research Design: Randomized, comparative-effectiveness study

Methodology /Technical Approach: A total of 225 patients with non-radicular chronic low back pain (LBP) with suspected facetogenic etiology will be randomized in a 2:2:1 ratio to one of 3 groups:

Group 1 will receive IA blocks with steroids and LA Group 2 will receive MBB with steroids and LA Group 3 will receive MBB with only saline

Those individuals who obtain significant (≥ 50% in groups 1 and 2,3) but temporary (< 1-month) relief will undergo radiofrequency (RF) denervation at their 1-month follow-up. In group 3, those patients who do not experience pain relief at 1-month will undergo RF denervation regardless of the pain relief they experience (as many practitioners in the military and civilian practices do without diagnostic blocks).1-3 Participants in Groups 1 and 2 who experience prolonged relief from their diagnostic/ therapeutic blocks with LA and steroids will not undergo RF denervation until their pain returns. Those individuals who experience prolonged relief lasting > 6 months will be given the option of repeating the diagnostic/ therapeutic block. In Groups 1, 2 and 3 patients who experience prolonged relief from the diagnostic blocks, follow-up visits will be at 1-month, 3-months and 6-months after the block, or until their pain relief wears off. In those who undergo denervation based on a positive block, follow-ups will be performed 1, 3 and 6-months after the denervation provided they continue to experience significant (> 50%) relief at each follow-up. Those individuals who fail to experience significant relief after denervation will be unblinded and exit the study per protocol.

DETAILED DESCRIPTION:
Two hundred and twenty five patients with suspected lumbar facet arthropathy scheduled to undergo diagnostic lumbar facet blocks will be enrolled in this study at WRNMMC and randomized in a 2:2:1 ratio into one of 3 groups. Group 1 will receive IA blocks with steroids and LA, group 2 will receive MBB with steroids and LA, and group 3 will receive MBB with only saline. Subjects and (but not injecting physicians) evaluators will be blinded throughout their participation in the study as to treatment allocation. The nerves and joints to be blocked will be determined by physical exam (i.e. the location of paraspinal tenderness), and radiological findings.

Group 1: The 80 patients in this group will undergo IA blocks under fluoroscopic guidance with 0.5 mL solutions containing a 50:50 mixture of 0.5% bupivacaine and 10 mg depomethylprednisolone (called "steroid"). In all cases, correct positioning will be confirmed by the administration of contrast. After the block, they will be administered a pain diary to maintain for the next 6 hours. In accordance with standard care, a positive response will be > 50% pain relief lasting at least 3 hours. Patients who have not undergone physical therapy (PT) will be sent for PT . The first follow-up will be at 1-month. In those individuals with a positive block whose pain has returned to baseline, RF denervation will be performed at the same levels done for the diagnostic block. Once adequate sensory stimulation is confirmed, a 1 mL mixture containing equal amounts of 2% lidocaine 0.5 mL) and 20 mg depo-methylprednisolone (0.5 mL) will be injected to reduce procedure-related pain and decrease the incidence of neuritis. For those patients who have persistent (> 50%) pain relief at 1-month, they will return for their 2nd follow-up at 3-months. If their pain relief persists at this point, their final follow-up will be 6-months post-procedure. Pain relief in this group that lasts > 6 months can be treated with repeat IA injections if the patient so desires, while that which persists for < 6 months will be treated with RF denervation. Patients who experience a negative diagnostic block, or who fail to obtain significant pain relief at any follow-up from their RF denervation, will exit the study per protocol to pursue alternative treatments

Group 2: The 80 patients in this group will undergo MBB blocks under fluoroscopic guidance with 0.5 mL solutions containing a 50:50 mixture of 0.5% bupivacaine and 10 mg of depo-methylprednisolone steroid. After the block, they will be administered a pain diary to maintain for the next 6 hours. Patients who have not undergone physical therapy will be sent for a PT program. The first follow-up will be at 1-month. In those individuals who do not experience significant pain relief, RF denervation will be performed at the same levels done for the diagnostic block, as described in 'Group 1'. For those patients who have persistent (> 50%) pain relief at 1-month, they will return for their 2nd follow-up at 3-months. If their pain relief persists at this point, their final follow-up will be 6-months post-procedure. Pain relief in this group that lasts > 6 months can be treated with repeat MBB if they desire, while that which persists for < 6 months will be treated with RF denervation. Patients who experience a negative diagnostic block, or who fail to obtain significant pain relief at any follow-up from their RF denervation, will exit the study per protocol to pursue alternative treatments.

Group 3: The 40 patients in this group will undergo IA blocks under fluoroscopic guidance with 0.5 mL of normal saline. After the block, they will be administered a pain diary to maintain for the next 6 hours. Patients who have not undergone physical therapy will be sent for PT. The first follow-up will be at 1-month. In those individuals who fail to experience significant pain relief at this time point, RF denervation will be performed at the same levels done for the diagnostic block, as described in 'Group 1'. For those patients who have persistent (> 50%) pain relief at 1-month, they will return for their 2nd follow-up at 3-months. If their pain relief persists at this point, their final follow-up will be 6-months post-procedure. Pain relief from the block in this group that lasts > 6 months can be treated with repeat MBB, while that which persists for < 6 months will be treated with RF denervation. In patients who do not experience significant pain relief at their 1-month follow-up, RF denervation will be performed. Those who experience a negative outcome from RF denervation, will exit the study per protocol to pursue alternative treatments.

During follow visits, subjects who have difficulty arranging for transportation can elect to conduct their follow-up visits over the telephone, via fax, or by e-mail, whichever is most convenient.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Suspected lumbar facet arthropathy based on history and physical exam (e.g. axial lower back pain, paraspinal tenderness, no pain referral below the knee)
* NRS back pain score > 4;
* MRI evidence of spinal pathology consistent with symptoms.

Exclusion Criteria:

* Untreated coagulopathy
* No MRI study
* Signs or symptoms of cauda equina syndrome
* Focal neurological signs and symptoms
* Allergic reactions to local anesthetics or contrast dye
* Serious medical or condition that might preclude optimal outcome
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Pain Score | 1 month
  0-10 numerical rating scale (NRS) average pain score after facet injection
Pain Score | 3 months
  0-10 numerical rating scale pain score after radiofrequency ablation

SECONDARY OUTCOMES:
Successful outcome after RF denervation | 1 month
  Proportion of patients in each arm who undergo RF denervation who experience a > 50% decrease in pain score and a satisfaction score > 3
Successful outcome after RF denervation | 3 months
  Proportion of patients in each arm who undergo RF denervation who experience a > 50% decrease in pain score and a satisfaction score > 3
Successful outcome after RF denervation | 6 months
  Proportion of patients in each arm who undergo RF denervation who experience a > 50% decrease in pain score and a satisfaction score > 3
Successful outcome after facet block | 1 month
  Proportion of patients in each arm who undergo RF denervation who experience a > 50% decrease in pain score and a satisfaction score > 3
Successful outcome after facet block | 3 months
  Proportion of patients in each arm who undergo RF denervation who experience a > 50% decrease in pain score and a satisfaction score > 3
Successful outcome after facet block | 6 months
  Proportion of patients in each arm who undergo RF denervation who experience a > 50% decrease in pain score and a satisfaction score > 3
Proportion of people with a positive pain diary | 1-day after injection
  Proportion of people who experience > 50% pain relief after the diagnostic block
Pain score | 1 month
  Worst NRS pain score 1 month after initial injection
Pain score | 3 months
  Average NRS pain score 3 months after initial injection
Pain score | 3 months
  Worst NRS pain score 3 months after initial injection
Pain score | 6 months
  Average NRS pain score 6 months after initial injection
Pain score | 6 months
  Worst NRS pain score 6 months after initial injection
Pain score | 1 month
  Average NRS pain score 1 month after RF denervation
Pain score | 1 month
  Worst NRS pain score 1 month after RF denervation
Pain score | 3 months
  Worst NRS pain score 3 months after RF denervation
Pain score | 6 months
  Average NRS pain score 6 months after RF denervation
Pain score | 6 months
  Worst NRS pain score 6 months after RF denervation
Function | 1 month
  Oswestry disability index score 1-month after initial injection
Function | 3 months
  Oswestry disability score 3-months after initial injection
Function | 3 months
  Oswestry disability score 6-months after initial injection
Function | 1 month
  Oswestry disability score 1-month after RF denervation
Function | 3 months
  Oswestry disability score 3-months after RF denervation
Function | 6 months
  Oswestry disability score 6-months after RF denervation
Satisfaction | 1-month
  Satisfaction on 1-5 scale 1-month after initial injection
Satisfaction | 3-months
  Satisfaction on 1-5 scale 3-months after initial injection
Satisfaction | 6-months
  Satisfaction on 1-5 scale 6-months after initial injection
Satisfaction | 1-month
  Satisfaction on 1-5 scale 1-month after RF denervation
Satisfaction | 3-months
  Satisfaction on 1-5 scale 3-months after RF denervation
Satisfaction | 6-months
  Satisfaction on 1-5 scale 6-months after RF denervation

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Cohen, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen SP, Huang JH, Brummett C. Facet joint pain--advances in patient selection and treatment. Nat Rev Rheumatol. 2013 Feb;9(2):101-16. doi: 10.1038/nrrheum.2012.198. Epub 2012 Nov 20. PMID 23165358
- [Background] Cohen SP, Raja SN. Pathogenesis, diagnosis, and treatment of lumbar zygapophysial (facet) joint pain. Anesthesiology. 2007 Mar;106(3):591-614. doi: 10.1097/00000542-200703000-00024. PMID 17325518
- [Derived] Cohen SP, Doshi TL, Constantinescu OC, Zhao Z, Kurihara C, Larkin TM, Griffith SR, Jacobs MB, Kroski WJ, Dawson TC, Fowler IM, White RL, Verdun AJ, Jamison DE, Anderson-White M, Shank SE, Pasquina PF. Effectiveness of Lumbar Facet Joint Blocks and Predictive Value before Radiofrequency Denervation: The Facet Treatment Study (FACTS), a Randomized, Controlled Clinical Trial. Anesthesiology. 2018 Sep;129(3):517-535. doi: 10.1097/ALN.0000000000002274. PMID 29847426